CLINICAL TRIAL: NCT04624308
Title: Toripalimab Plus TPF Inductive Chemotherapy and Definitive Radiotherapy for Resectable Locally Advanced Hypopharyngeal Squamous Cell Carcinoma, Efficacy and Safety: a Phase II Prospective Cohort Study
Brief Title: Toripalimab Plus TPF Chemotherapy and Radiotherapy for LA-HPSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yan (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor-Investigator, Sun Yan, Principal Investigator, Chief of Head and Heck Group of Radiotherapy Department, Peking University Cancer Hospital, Peking University, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-JS001-HPSCC
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Hypopharyngeal Neoplasm Malignant Primary
Keywords: hypopharyngeal carcinoma; radiotherapy; inductive chemotherapy; PD-1 inhibitor
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPF inductive chemotherapy plus Toripalimab and radiotherapy plus Toripalimab (Experimental): TPF inductive chemotherapy plus Toripalimab for 3 cycles, and radiotherapy plus Toripalimab if the inductive treatment efficacy is CR or >75%PR. If not, operation is suggested.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg d1，Q3W. Given with TPF during inductive chemotherapy and definitive radiotherapy.
  Other Names: Tuoyi

SUMMARY:
TPF is the standard regime of inductive chemotherapy for squamous carcinoma of head and neck. If the primary tumor shrinks obviously (complete remission or >75% partial remission )after inductive chemotherapy, CCRT is suggested as the definitive therapy, for the tumor is sensitive to chemotherapy. If the primary tumor shrinks a little or progresses after inductive chemotherapy, operation is suggested as the definitive therapy to get a longer survival.

DETAILED DESCRIPTION:
Inductive chemotherapy plus CCRT or operation is an option of organ preservation for patients of hypopharyngeal carcinoma. Many clinical studies have demonstrated that inductive chemotherapy plus CCRT achieved the same prognosis as total laryngectomy, and minimized the damage of normal tissue. TPF is the standard regime of inductive chemotherapy for squamous carcinoma of head and neck. If the primary tumor shrinks obviously (complete remission or >75% partial remission )after inductive chemotherapy, CCRT is suggested as the definitive therapy, for the tumor is sensitive to chemotherapy. If the primary tumor shrinks a little or progresses after inductive chemotherapy, operation is suggested as the definitive therapy to get a longer survival. This is a prospective, phase II, cohort study. We designate TPF plus Toripalimab as the inductive regime, expecting a higher complete remission rate and longer PFS and OS. And we replace the CCRT with radiation plus Toripalimab to decrease the adverse events of CCRT.

ELIGIBILITY:
Inclusion Criteria:

1. 18y ≤age≤65y;
2. ECOG：0-1；
3. Histology：squamous cell carcinoma, located in hypopharynx;
4. clinical stage: cT1N1-3M0、cT2-3N0-3M0，organ-preservation-intent regime is made after multidisciplinary treatment(MDT) discussion. Efficacy evaluation will be made according to RECIST 1.1 after inductive chemotherapy, and the following treatment will be chosen according to the results of efficacy evaluation.
5. never received any previous treatment, including radiotherapy, chemotherapy, or immune therapy, et al.
6. at least one measurable lesion (RECIST 1.1 criteria).
7. expected survival ≥6 months.
8. no contraindications of radiotherapy, chemotherapy and immune therapy.
9. functions of main organs A. WBC≥3.0x109 /L，ANC≥1.5x109/L B. HB≥90g/L C. PLT≥100x109 /L D. serum albumin≥2.8g/dL E. TBil ≤1.5xULN，ALT、AST≤3.0xULN F. serum creatinine ≤1.5xULN or creatinine clearance rate>60mL/min（Cockcroft-Gault） G. APTT and INR ≤1.5xULN
10. contraception
11. voluntary and compliance.

Exclusion Criteria:

1. other histology cancers located in hypopharynx.
2. synchronous or metachronous cancers located in other sites.
3. allergy to monoclonal antibody.
4. uncontrollable heart disease or symptoms.
5. uncontrollable infections.
6. fever of unknown origin>38.5℃ during screening or before administration.
7. active autoimmune disease.
8. history of immunodeficiency disorders, including HIV.
9. active HBV or HCV.
10. history of interstitial lung disease.
11. active tuberculosis.
12. received any drugs listed below: A. received any study drug 4 weeks before first dose of Toripalimab. B. received any anti-cancer drug 4 weeks before first dose of Toripalimab. C. received any glucocorticoids （>10mg prednison per day） 2 weeks before first dose of Toripalimab.

    D. received any cancer vaccine 4 weeks before first dose of Toripalimab. E. received any operation or trauma 4 weeks before first dose of Toripalimab. F. recruited in other study.
13. uncontrollable hypertension.
14. uncontrollable type 2 diabetes；
15. hemorrhagic tendency.
16. drug or alcoholic abuse.
17. woman during pregnancy or lactation period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 3 months after treatment
  Complete remission rate 3 months after treatment

SECONDARY OUTCOMES:
ORR | 3 months after treatment
  objective response rate
DCR | 5 year
  disease control rate
PFS | 5 year
  progression free survival
OS | 5 year
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data is administered by Peking University Cancer Hospital, the investigators need to request related department for sharing IPD.